CLINICAL TRIAL: NCT01934985
Title: Dynamic Cardiac SPECT Imaging
Acronym: SPECT
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Lawrence Berkeley National Laboratory (LBNL) (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 5R01HL050663 (NIH); 5R01HL050663 (NIH)
Record Dates: First submitted 2013-08-19; First posted 2013-09-04 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Disease
Keywords: Single-Photon Emission-Computed Tomography; Myocardial Perfusion Imaging; Ischemia; Stress test; Coronary Artery Disease (CAD); Coronary Flow Reserve (CFR); Coronary Angiography
MeSH Terms: conditions — Coronary Artery Disease; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1: Patients scheduled to have clinically indicated stress MPI with low pre-test likelihood (0-15%) of coronary disease based on criteria of Diamond and Forrester. And those who have already had a clinical indicated stress MPI in the last three years with a low likelihood of having active coronary disease with no significantly narrowed coronary arteries.
- Group II: Patients in Group II who will have the dynamic imaging protocol studies after SCA, patients will be selected for protocol enlistment only if the decision is made by the patient's physician, based totally on clinical and social factors, that any considered revascularization intervention would not be performed on the day of diagnostic selective coronary angiography (SCA) and will be performed electively, at least 4 to 7 days later. Viability will be assessed in these patients only in the presence of WM abnormalities, and with serial analysis of WM, as described above. Patients will be followed for death or infarction or other events more than 3 months after study, for up to 3 years following participation in the protocol.
- Group III: Patients found at SCA to have lesions of "borderline" clinical significance, preferably in the absence of other associated lesions.
- Group IV: Patients who were diagnosed with advanced heart failure including patients who had or will have cardiac resynchonization therapy (CRT) or a heart transplant.

SUMMARY:
The investigators propose a 4 year prospective, observational study of 40 patients yearly, comparing conventional clinically indicated SPECT and PET perfusion with dynamic rest/stress MPI studies with coronary angiography, in some cases performed with quantitative coronary anatomy and flow as well as quantitative 13N-ammonia PET MPI. Methods will also be assessed for their ability to determine myocardial viability by comparing regional wall motion (WM) on clinically indicated serial ventriculography, echocardiography or gated SPECT MPI in those protocol patients with WM abnormalities who subsequently undergo revascularization. Patient studies will begin in the first study year based on those methods already developed and integrate new advances as they become evident.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had clinically indicated stress MPI with a low pre-test likelihood (0 - 15% ) of coronary disease based on the criteria of Diamond and Forrester.
* Patients who have already had a clinically indicated stress MPI in the last three years with a low likelihood of having active coronary disease with no significantly narrowed coronary arteries.
* Patients whose clinically indicated stress MPI demonstrates clear abnormalities and who are likely to go on to SCA for clinical indications.
* If, after conventional and dynamic MPI some of these patients do not have SCA, they will still be followed for events for up to 3 years following participation in the protocol. To avoid delays and unnecessary procedures among patients in Group II who will have the dynamic imaging protocol studies after SCA, patients will be selected for protocol enlistment only if the decision is made by the patient's physician, based totally on clinical and social factors, that any considered revascularization intervention would not be performed on the day of diagnostic SCA and will be performed electively, at least 4 to 7 days later.
* Patients found at SCA to have lesions of "borderline" clinical significance, preferably in the absence of other associated lesions.

Exclusion Criteria:

* Cannot give informed consent
* Unable or unwilling to return for a second stress imaging study
* Cannot cooperate for adequate SPECT or PET supine and/or prone imaging
* Pregnant females
* Patients under 21 years old
* Active bronchospasm - No theophylline for 48 hours prior to study
* Heart block more severe than Wenckebach block
* Patients with uncomplicated infarction will not be included if they cannot have an exercise test later than 8 weeks of the event or a vasodilator pharmacologic stress test at least 24 hours or more after the event
* Coronary bypass surgery within 8 weeks
* Symptoms of congestive heart failure at rest
* Has had an event or change in drug regimen since the initial stress test.
* Has serious response to or side effect from initial clinical stress test induced ST elevation, hypotension, prolonged arrhythmia, bronchospasm.
* Has had a clinical event since last coronary angiogram, angioplasty, or coronary surgery.
* Has had 201Tl rest SPECT MPI prior to dynamic imaging

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University of California, San Francisco (UCSF) Cardiology Clinics
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Coronary Flow Reserve | Length of procedure- 90 min
  The coronary flow reserve will be measured by comparing the rest and stress exams on the dynamic SPECT scans using developed algorithms. The accuracy will be compared with clinical PET, coronary angiography, and clinical SPECT.

CONTACTS AND LOCATIONS:
Overall Officials: Youngho Seo, Phd, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco Imaging Center, San Francisco, California, United States